CLINICAL TRIAL: NCT05796024
Title: Derivation and Validation of a National Multicenter In-hospital Mortality Risk Stratification Model - the Ex-Care Model II
Brief Title: Derivation and Validation of the Extended Care (Ex-Care) Model II
Acronym: Ex-CareII
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.0192
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Complications
Keywords: risk assessement; validation study; postoperative; mortality
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation Cohort: The derivation cohort will correspond to approximately 70% of the total sample to be analyzed in the study. The Ex-Care II risk model will build upon it. It is composed of patients operated in the participating institutions.
- Validation Cohort: Composed of the remaining 30% of the sample. It will be used for the external validation of the Ex-Care II model

SUMMARY:
The goal of this study is to develop a novel surgical risk stratification tool designed to adults operated in Brazil. The main question it aims to answer is:

•Is the Extended Care (Ex-Care) II model a good tool to assess the risk of death among patients operated in Brazilian hospitals within 30 days after surgery?

Information of patients undergoing surgery in the participating hospitals over a period of 24 months will be analyzed to evaluate the relationship of some patients characteristics (called predictors) with the study outcome (probability of death).

The sample will be divided in two groups. The first, called derivation sample, will be used for the development of the Ex-Care II model. The second, called validation sample, will evaluate the performance of this new model.

DETAILED DESCRIPTION:
From four predictors collected preoperatively ( American Society of Anesthesiology Physical Status (ASA-PS) classification, age, extent of surgery and its nature - elective vs urgency/emergency), through a multilevel logistic regression, a post-surgical in-hospital mortality prediction model will be developed, the Ex-Care II model. Discrimination and calibration measures will be used to determine the accuracy of the model. In addition, each predictor will have their odds ratio calculated for the study outcome. Once this model is developed, it will have its external validity tested in a second sample, using the same accuracy metrics.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 16 years of age undergoing elective, urgent or emergency surgeries in the hospitals participating in the study

Exclusion Criteria:

* Diagnostic procedures, with sedation only or with local anesthesia
* Patients undergoing liver, pulmonary and/or cardiac transplant surgery, as well as those diagnosed with brain death submitted to organ donation
* In the event that the patient undergoes more than one surgical intervention in the same hospitalization, only the major procedure will be considered for the purpose of denouement

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 16 years or older undergoing surgery in hospitals in different regions of Brazil
Sampling Method: Non-Probability Sample
Enrollment: 107372 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Develop and validate a model for predicting the risk of in-hospital death within 30 days postoperatively, from a sample composed of patients operated in Brazil | Surgery day up to 30 days postoperatively
  From four predictors collected preoperatively, the developed model will be able to estimate the probability of in-hospital death of patients undergoing surgery in Brazilian hospitals. For the creation of this tool, multilevel logistic regression will be made with hospital as a random effect

SECONDARY OUTCOMES:
Develop smartphone application contemplating the new model developed | Preoperative
  In order to facilitate the use of the Ex-Care II model by health professionals involved in perioperative care, it will be created and made available on the main platforms for smartphones application that will allow the measurement of surgical risk by this new tool.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana C Stefani, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Passos SC, Stahlschmidt A, Blanco J, Spader ML, Brandao RB, Castro SMJ, Gutierrez CS, Silva Neto PCD, Stefani LPC. Derivation and validation of a national multicenter mortality risk stratification model - the ExCare model: a study protocol. Braz J Anesthesiol. 2022 May-Jun;72(3):316-321. doi: 10.1016/j.bjane.2021.07.003. Epub 2021 Jul 26. PMID 34324938
- [Derived] Passos SC, de Jezus Castro SM, Stahlschmidt A, da Silva Neto PC, Irigon Pereira PJ, da Cunha Leal P, Lopes MB, Dos Reis Falcao LF, de Azevedo VLF, Lineburger EB, Mendes FF, Vilela RM, de Araujo Azi LMT, Antunes FD, Braz LG, Stefani LC. Development and validation of the Ex-Care BR model: a multicentre initiative for identifying Brazilian surgical patients at risk of 30-day in-hospital mortality. Br J Anaesth. 2024 Jul;133(1):125-134. doi: 10.1016/j.bja.2024.04.001. Epub 2024 May 10. PMID 38729814